CLINICAL TRIAL: NCT04026295
Title: Short-Burst Interval Treadmill Training to Improve Community Walking Activity and Mobility in Cerebral Palsy
Brief Title: Short-Burst Interval Treadmill Training Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kristie Bjornson (Other)
Collaborators: University of Washington (Other); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor-Investigator, Kristie Bjornson, Professor, Pediatrics, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD098270 (NIH)
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy
Keywords: treadmill training; gait; short burst interval locomotor training; spastic
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either short-burst interval locomotor treadmill training (SBLTT) or traditional locomotor treadmill training (TLTT)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short burst Interval Treadmill Training (SBLTT) (Experimental): SBLTT will consist of short-bursts (30 seconds) of high speed walking alternating with 30 seconds of low/moderate speed walking. Participant will receive 40 home-based sessions (5x/week for 8 weeks) of SBLTT
  Interventions: Behavioral: Short Burst Interval Treadmill Training (SBLTT)
- Traditional Locomotor Treadmill Training (TLTT) (Active Comparator): TLTT will consist of walking at steady-state speeds. Participant will receive 40 home-based sessions (5x/week for 8 weeks) of TLTT
  Interventions: Behavioral: Traditional Locomotor Treadmill Training (TLTT)

INTERVENTIONS:
Behavioral: Short Burst Interval Treadmill Training (SBLTT) — SBLTT will consist of short-bursts (30 seconds) of high speed walking alternating with 30 seconds of low/moderate speed walking. Total duration of walking per session will be up to 30 minutes of the 30 second alternating intervals (30sec high / 30sec low/moderate) with rests as needed. Both groups will receive 40 sessions delivered 5x/week for 8 weeks. Initial speeds for high speed walking will be 75-80% of each participant's over ground baseline fast walking speed, and low/moderate speed will be 75-80% of self-selected speed calculated from the 10-Meter Walk Test.
  Arms: Short burst Interval Treadmill Training (SBLTT)
Behavioral: Traditional Locomotor Treadmill Training (TLTT) — TLTT group will receive the same number of sessions (40) delivered 5x/week for 8 weeks with a total duration of walking per session up to 30 minutes with rests as needed. TLTT will consist of walking at steady-state speeds. Initial treadmill speed will be 75-80% of over ground self-selected walking speed. The overall goal will be to achieve 30 minutes of walking at a steady-state walking speed within each session. Speed will be increased on the next session by .1 to .4mph when the subject can walk for 30 minutes on the treadmill at the current speed with an OMNI score of < 6/10.
  Arms: Traditional Locomotor Treadmill Training (TLTT)

SUMMARY:
Ambulatory children with cerebral palsy (CP) walk predominately in low intensity stride rates with little variability, thus limiting their walking activity and ability to participate in daily life. In contrast, typically developing (TD) children engage in short bursts of intense walking activity interspersed with varying intervals of low intensity walking within daily life. In order to optimize motor learning, active participation, task-specific training and multiple repetitions or massed practice is required to learn new motor skills. Short bursts of vigorous intensity locomotor treadmill training (SBLTT) alternating with low/moderate intensity was specifically designed to mimic activity patterns of TD children in a massed practice format. Pilot data suggests that SBLTT is feasible and enhances walking capacity and performance in daily life for children with CP. This project will examine the effect of SBLTT versus an equivalent dosage of traditional locomotor treadmill training (TLTT) on the primary outcomes of walking capacity and performance in children with CP and whether the effects of SBLTT on walking capacity and performance are mediated by improvements in in muscle power generation. The scientific premise is that SBLTT, that approximates the walking intensity patterns of typically developing (TD) children through a home-based massed practice protocol, will be more effective than TLTT in improving walking capacity and performance. We hypothesize that SBLTT strategies for children with CP modeled on walking patterns of TD children, will be positively mediated by muscle power generation and subsequently improve walking capacity and community walking performance and mobility. Specific aims. Aim #1. Determine the immediate and retention effects of short-burst interval LTT (SBLTT) on walking capacity in ambulatory children with CP. Aim #2. Examine the effects of treatment on community-based walking activity performance and mobility. Aim #3. Explore whether the effects of SBLTT on walking capacity and performance are mediated by muscle power generation. The proposed research will be the first step in a continuum of research that is expected to direct locomotor training protocols and rehab strategies across pediatric disabilities and positively effecting the community walking performance and mobility for children with CP.

DETAILED DESCRIPTION:
In a randomized clinical trial, 72 ambulatory children with spastic CP (6-10 yrs.) will receive either SBLTT or an equivalent dosage of TLTT for 40 sessions, 5x/week for 8 weeks in a massed practice format. The only difference between training protocols will be the variable training (interval fast versus steady state walking speeds). Thus, the key ingredient will be the intensity of the interval training delivered in a serial blocked practice schedule. Outcomes will be collected at baseline, 4 and 8 weeks to assess dosage, and 24 weeks post training for long term retention with the primary endpoint at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral and unilateral spastic cerebral palsy
* Gross Motor Function Classification Levels II & III
* Ages 6 years to < 11 years

Exclusion Criteria:

* Orthopedic or neurosurgery < 9 months prior
* Injection therapy (Botulinum Toxin/Phenol) < 3 months prior

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Walking Capacity-Self-selected walking speed | Baseline to 8 weeks
  10 Meter Walk Test
Walking Capacity-Fast walking speed | Baseline to 8 weeks
  10 Meter Walk Test- fast speed
Walking Capacity-Endurance | Baseline to 8 weeks
  One Minute Walk Test
Walking Performance-level | Baseline to 8 weeks
  StepWatch (SW) accelerometry - average total steps per day
Walking Performance-Intensity | Baseline to 8 weeks
  StepWatch (SW) accelerometry - percent of strides/day in medium/high stride rates.
Knee extensor muscle power | Baseline to 8 weeks.
  Isokinetic Average Power for Knee extensors at 60deg/s as measured by Biodex.

SECONDARY OUTCOMES:
Walking Mobility -level home | Baseline to 8 weeks
  StepWatch (SW) synchronized with Global Positioning System (GPS) home setting- average strides per day.
Walking Mobility-intensity home | Baseline to 8 weeks
  StepWatch (SW) synchronized with Global Positioning System (GPS) home setting- percent average strides/day in medium/high stride rates.
Mobility-Patient Reported Outcome | Baseline to 8 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS v1.0 Parent Pediatric Profile) Mobility domain score
Family Gait Priorities and Quality of gait | Baseline to 8 weeks
  Parent report Gait Outcome Assessment List (GOAL).total score
Knee extensor muscle torque | Baseline to 8 weeks.
  Isokinetic Peak Torque for knee extensors at 60 deg/s as measured by Biodex.
Walking Mobility-intensity community | Baseline to 8 weeks
  StepWatch (SW) synchronized with Global Positioning System (GPS) community setting- percent average strides/day in medium/high stride rates.
Walking Mobility -level community | Baseline to 8 weeks
  StepWatch (SW) synchronized with Global Positioning System (GPS) community setting- average strides/day.

CONTACTS AND LOCATIONS:
Overall Officials: Kristie F Bjornson, PhD, PT, Principal Investigator — Seattle Children's Hospital; Noelle Moreau, PhD, PT, Principal Investigator — Lousianna State University in New Orleans
Locations (2):
- United States (2):
  - Lousianna State University Health Sciences Center New Orleans, New Orleans, Louisiana
  - Seattle Childrens Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No